CLINICAL TRIAL: NCT04571229
Title: Expanded Access Use of L-MTP-PE for the Treatment of Osteosarcoma
Status: Available | Type: Expanded Access
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-324
Record Dates: First submitted 2020-09-16; First posted 2020-09-30 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Osteosarcoma
Keywords: L-MTP-PE; Expanded Access; 20-324
MeSH Terms: conditions — Osteosarcoma | interventions — mifamurtide

INTERVENTIONS:
Drug: L-MTP-PE — L-MTP-PE will be administered at a dose of 2mg/m2 (maximum dose 4 mg), twice weekly for 12 weeks and weekly for an additional 24 weeks, for a total of 48 doses in 36 weeks.

SUMMARY:
This expanded access protocol will allow access to treatment with L-MTP-PE for people with osteosarcoma. L-MTP-PE is an investigational drug that has not been approved by the FDA to treat any condition, including osteosarcoma. L-MTP-PE works by activating certain types of white blood cells, and these active white blood cells help the immune system kill cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of osteosarcoma of any age Note: Patients with either newly diagnosed or relapsed osteosarcoma are eligible.
* Surgical resection or other definitive local control therapy of all clinically detectable sites of osteosarcoma
* L-MTP-PE is deemed to be of potential benefit by the treating investigator
* Willing and able to understand and sign informed consent and assent as appropriate
* Life expectancy > 6 weeks
* Adequate organ function as follows:
* Adequate bone marrow function defined as:

  * absolute neutrophil count (ANC) ≥ 750/mm^3
  * platelet count ≥ 30,000/ mm^3
  * hemoglobin ≥ 8 g/dl
* Adequate renal function defined as:

  * Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min/1.73m^2 OR
  * Serum creatinine ≤ 2x the upper limit of normal based on age/gender
* Adequate liver function defined as:

  * Bilirubin (sum of conjugated + unconjugated) ≤ 2x upper limit of normal for age or ≤ 4x upper limit of normal if thought to have Gilbert's disease
  * AST or ALT ≤ 3x upper limit of normal or ≤ 5x upper limit of normal for patients with liver metastases
* Willing to use a barrier method of contraception throughout the course of the study and for 1 year after participation if relevant

Exclusion Criteria:

* Use of chronic steroids of other immunosuppressive agents
* Pregnant or breast feeding

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slotkin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm